CLINICAL TRIAL: NCT00666900
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Dose-Ranging Study to Evaluate IDP-107 Versus Placebo in the Treatment of Severe Acne Vulgaris With Nodules
Brief Title: A Clinical Study Evaluating the Safety and Efficacy of IDP-107 in Patients With Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dow Pharmaceutical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DPSI-IDP-107-P2-01
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Low Strength IDP-107
- 2 (Experimental)
  Interventions: Drug: High Strength IDP-107
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Low Strength IDP-107 — Once a day for 12 weeks
  Arms: 1
Drug: High Strength IDP-107 — Once a day for 12 weeks
  Arms: 2
Drug: Placebo Comparator — Once a day for 12 weeks
  Arms: 3

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of IDP-107 in treating patients with acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Presence of inflammatory and non-inflammatory lesions

Exclusion Criteria:

* Dermatological conditions of the face that could interfere with clinical evaluations
* Female subjects who are pregnant, nursing, planning a pregnancy, or become pregnant during the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the number of inflammatory lesions | 12 weeks
Improvement from baseline in global severity | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in the number of non-inflammatory lesions | 12 weeks

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Dermatology Research of Arkansas, PLLC, Little Rock, Arkansas
  - RADY Children's Hospital - San Diego, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - Solano Clinical Research, Vallejo, California
  - Cherry Creek Research, Inc., Denver, Colorado
  - FXM Research Corp., Miami, Florida
  - Michigan Center for Skin Care Research, Clinton Township, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Skin Specialist, PC, Omaha, Nebraska
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Dermatology Associates of Rochester, Rochester, New York
  - DermResearchCenter of New York, Inc., Stony Brook, New York
  - University of North Carolina Hospitals and School of Medicine, Chapel Hill, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Arlington Research Center, Inc., Arlington, Texas
  - DermResearch, Inc., Austin, Texas
  - J & S Studies, Inc., Bryan, Texas
  - The Center for Skin Research, Houston, Texas
  - South Valley Dermatology, West Jordan, Utah
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Premier Clinical Research, Spokane, Washington
  - Madison Skin & Research, Inc., Madison, Wisconsin